CLINICAL TRIAL: NCT04110158
Title: A Study on Chronic Constipation Etiology and Risk Factors Among School Age Children in Assuit University Children Hospital
Brief Title: Chronic Constipation in Children Among School Children is Assuit University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Mohamed Hussien, FAmhussien, Assiut University
Other Study IDs: Chronic constipation
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Chronic Constipation in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the work to show rate of constipation among school age children in Assuit University Children Hospital

DETAILED DESCRIPTION:
Childhood constipation is a frequently overlooked global health problem, which is developing in a public health issue in many parts of the world.(1) Constipation is one of the commonest digestive complaints in children(2) Constipation has long been considered a symptom, rather than a disease(3)

It is often perceived as infrequent motions or passage of hard stools. Some defined constipation as less than 3 bowel motions per week)4(

or as difficulty in passing stools (5) Approximately 0.5% of school children have defecation frequency less than 3 per week and 0.3% have fecal incontinence(6) Furthermore, 20% of children also have at least 1 clinical feature of constipation.7 Therefore, it is important to use diagnostic criteria based on multiple symptoms to define constipation

ELIGIBILITY:
Inclusion Criteria:school age children 4:18 years old -

Exclusion Criteria: neonates and younger than 4years children

-

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children between 4:18 years old complain of constipation for a period long than 2 months
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
A.study on chronic Constipation Etiology and risk factors among school age children in Assuit University Children Hospital | Baseline
  Constipation, risk factors ,management and outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Tawfeek, Study Director — Mustafa.tawfeek1@med.au.edu.eg

REFERENCES:
- [Background] Rajindrajith S, Devanarayana NM. Constipation in children: novel insight into epidemiology, pathophysiology and management. J Neurogastroenterol Motil. 2011 Jan;17(1):35-47. doi: 10.5056/jnm.2011.17.1.35. Epub 2011 Jan 26. PMID 21369490